CLINICAL TRIAL: NCT00183599
Title: Effect of Type and Duration of Therapy on Treatment for Gambling
Brief Title: Gambling and Brief Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Donaghue Medical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-205; DF#00-121
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Gambling
Keywords: Brief interventions; Motivational Enhancement Therapy; Cognitive Behavioral Therapy
MeSH Terms: conditions — Gambling | interventions — Motivational Interviewing; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Behavioral: 5 Minutes of Simple Advice
- 2 (Experimental)
  Interventions: Behavioral: Motivational Enhancement Therapy (MET)
- 3 (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: 5 Minutes of Simple Advice
  Arms: 1
Behavioral: Motivational Enhancement Therapy (MET)
  Arms: 2
Behavioral: Cognitive Behavioral Therapy (CBT)
  Arms: 3

SUMMARY:
This study will compare four different combinations and durations of motivational enhancement therapy, cognitive behavioral therapy, and brief advice treatments for gambling versus a non-intervention condition to determine which is most effective in reducing problem gambling.

DETAILED DESCRIPTION:
Gambling, if done compulsively, can cause psychological, physical, social, and vocational problems. Problem gambling, or compulsive gambling, is a progressive addiction characterized by a preoccupation with gambling, a need to bet more money more frequently, restlessness or irritability when attempting to stop, and gambling more to make up for losses. This study will compare four different combinations and durations of motivational enhancement therapy (MET), cognitive behavioral therapy (CBT), and brief advice treatments for gambling versus a non-intervention condition to determine which is most effective in reducing problem gambling.

This open-label study will last a total of 9 months. Participants will be randomly assigned to one of four groups. Group 1 will have no intervention and will be instructed to call if they experience any gambling problems. Group 2 will receive 5 minutes of education on the hazards of heavy gambling. In addition, they will receive a 1-page brochure on problem gambling and its consequences. Group 3 will receive a 1-hour session of MET focused on increasing commitment to change by raising awareness of personal consequences of gambling. Group 4 will receive the same MET session as Group 3, as well as three 1-hour sessions of CBT focused on identifying specific social and mood cues associated with gambling. Treatment will end at Week 4. Participants will have two follow-up sessions held over the phone at Week 6 and again 9 months after enrollment. Gambling behavior, employment status, alcohol and drug use, psychiatric problems, and family problems will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for problem gambling
* Two or more gambling episodes per month for 2 months prior to enrollment
* Has spent at least $50 per month on gambling for 2 months prior to enrollment

Exclusion Criteria:

* Any uncontrolled psychiatric conditions
* Severe cognitive impairment
* Currently receiving treatment for gambling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 1999-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Addiction Severity Index (ASI)-gambling severity scores | measured at baseline, Week 6, and 9 months
Amount spent gambling | measured at baseline, Week 6, and 9 months
Days gambled | measured at baseline, Week 6, and 9 months
Proportion meeting problem gambling criteria | measured at baseline, Week 6, and 9 months
Proportion abstinent | measured at baseline, Week 6, and 9 months

SECONDARY OUTCOMES:
Psychosocial functioning | measured at baseline, Week 6, and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Petry, PhD, Principal Investigator — UConn Health
Locations (6):
- United States (6):
  - LMG, Bridgeport, Connecticut
  - University of Connecticut Health Center, Farmington, Connecticut
  - CSAC, Hartford, Connecticut
  - Southern CT State University, New Haven, Connecticut
  - LMG, Stamford, Connecticut
  - University of Connecticut, Storrs, Connecticut